CLINICAL TRIAL: NCT01375465
Title: The 001-DIOR Multicenter Registry (A Novel Percutaneous Coronary Intervention With the New Paclitaxel-eluting Balloon DIOR in Ostial Bifurcated Lesions)
Brief Title: The 001-DIOR Multicenter Registry
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eurocor GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eur-002
Record Dates: First submitted 2011-06-16; First posted 2011-06-17 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dior (Other): One arm observational registry using the Dior paclitaxel eluting balloon for the treatment of de novo ostial bifurcated lesions.
  Interventions: Device: DIOR drug-eluting PTCA balloon

INTERVENTIONS:
Device: DIOR drug-eluting PTCA balloon — Treatment for 45 seconds with the DIOR balloon (3 µg/mm2 Paclitaxel concentration on balloon surface)

SUMMARY:
The 001 DIOR study is a prospective, multicenter registry of percutaneous coronary intervention (PCI) to assess the clinical success, efficacy and safety of the Paclitaxel-eluting balloon DIOR (Eurocor GmbH, Germany) for the treatment of de novo ostial bifurcated lesions (001 of Medina classification). The DIOR balloon will be used to treat the stenotic site branch.

ELIGIBILITY:
Inclusion Criteria:

* De novo bifurcated lesions 001 of Medina classification, with significant stenosis only in the ostium of the side branch and a reference vessel diameter is bigger or equal 2.0mm; the DIOR balloon will be used to the treat the side branch.
* The patient has clinical evidence of myocardial ischemia (stable or unstable angina, acute and non acute myocardial infarction, silent ischemia: ECG, exercise test, etz...)
* As the maximal length of the DIORTM balloon is 30 mm, all eligible lesions should be no longer than 25 mm to ensure an adequate drug elution in the treated segment, avoiding the phenomenon of "geographical miss" .
* Target lesion(s) stenosis is more or equal 50% by visual estimation.

Exclusion Criteria:

* Cardiogenic shock
* Any serious disease that might limit patient survival to less than one year
* Inability to perform clinical follow-up for a period of 1 year
* Left main bifurcation lesions: ostial left circumflex or ostial left anterior descending artery stenosis.
* Lesion length > 25 mm
* Target vessel reference diameter < 2mm
* Stenosis < 50% of the reference luminal diameter
* Severe angiographic calcification at the level of the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-02; Primary Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events (MACE) | 6 months
  MACE rate defined as the rate of cardiac death and/or myocardial infarction (MI) and/or target lesion revascularization (TLR)

SECONDARY OUTCOMES:
target vessel revascularization (TVR) rate, either symptom or ischemia-driven | 6 months
Segment treated thrombosis (STT), according to ARC definitions | 6 months
Late Lumen Loss | 6 months
  Late lumen loss determinated by control angiography
Binary restenosis rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Serra, MD, PhD, Principal Investigator — Hospital Sant Pau, Barcelona; Beatriz Vaquerizo, MD, PhD, Principal Investigator — Hospital Sant Pau, Barcelona
Locations (3):
- Spain (3):
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Trías i Pujol, Barcelona